CLINICAL TRIAL: NCT03820765
Title: Analysis of Cessation of the Dialysis Treatment in Reinbek-Northern Germany
Brief Title: Cessation of Dialysis Treatment in Reinbek and Geesthacht
Acronym: CoDiRaG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Markus Meier, MD, Consultant Nephrologist Dialysis and Apheresis, University of Luebeck
Other Study IDs: CODIRAG-2019
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Complication of Renal Dialysis; Long-Term Disorder of Dialysis
Keywords: Hemodialyis, Peritonealdialysis, Qualitiy assurance dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, approximately 80.000 patients with end stage renal disease (ESRD) in Germany undergo chronic renal replacement therapy, either as hemodialysis or peritonealdialysis. Since the nationwide registry for chronic dialysis patients (QuasiNiere) was terminated in 2006, no data exist from that time on regarding alterations in morbidity and mortality of patients with end stage renal disease in Germany.

With this study we start a single center prospective registry of all patients undergoing hemodialysis or peritonealdialysis therapy in our two nephrology departments Reinbek and Geesthacht. In these centers we perform approximately 34.000 hemodialysis sessions and supervise about 10.000 peritoneal treatment days of about 300 ESRD patients annually.

The aim of the study is to analyze all patients who stopped dialysis treatment in our centers due to death, kidney transplantation, recovery of renal function or other causes. Patients characteristics such as underlying renal diseases, duration of dialysis, co-morbidities as well as laboratory parameters will be recorded.

The data is collected with an Microsoft Access Database and analyzed by a statistician of the University of Luebeck (Germany). Power calculations revealed, that at least 200 patients were necessary to detect differences in particular interesting variables such as vascular access or the need of palliative care. During the last years at least 50 patients stopped chronic renal replacement therapy at out centers annually. Thus, the first interims evaluation is expected after 4 years.

The results of our study are important to estimate the development of patient age and renal diseases responsible for dialysis therapy in our centers. Moreover, the results may add important information to our internal quality assurance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease and hemodialyis or peritonealdialysis
* Renal replacement therapy performed in our centers Reinbek or Geesthacht
* at least 4 weeks of dialysis treatment in any of our two treatment sites

Exclusion Criteria:

* dialysis treatment period in our centers shorten than 4 weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with the necessity of chronic renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Dialysis time (months) as a function of patient age (years). | 4 years
  Differences of the dialysis time (months) between patients < 65 years, 65-80 years and > 80 years.
Underlying renal disease of ESRD patients | 6 years
  Differences of the underlying renal disease between patients with initiation of dialysis prior to 31.12.2012 or after 1.1.2013

SECONDARY OUTCOMES:
Albumin concentration of ESRD patients | 6 years
  Serum albumin concentration of dialysis patients at initiation of treatment, after 6 months and at cessation of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Markus Meier, MD, Principal Investigator — University of Luebeck
Locations (1):
- Nephrology Center Reinbek and Geesthacht, Reinbek, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCullough K, Sharma P, Ali T, Khan I, Smith WC, MacLeod A, Black C. Measuring the population burden of chronic kidney disease: a systematic literature review of the estimated prevalence of impaired kidney function. Nephrol Dial Transplant. 2012 May;27(5):1812-21. doi: 10.1093/ndt/gfr547. Epub 2011 Sep 29. PMID 21965592
- [Result] Schober-Halstenberg HJ. End-stage renal disease in aging societies: a global perspective. J Ren Nutr. 2009 Sep;19(5 Suppl):S3-4. doi: 10.1053/j.jrn.2009.06.015. No abstract available. PMID 19712874
- [Result] Frei U, Schober-Halstenberg HJ. Annual Report of the German Renal Registry 1998. QuaSi-Niere Task Group for Quality Assurance in Renal Replacement Therapy. Nephrol Dial Transplant. 1999 May;14(5):1085-90. doi: 10.1093/ndt/14.5.1085. PMID 10344342
- [Result] Frei U. Quality assurance in renal replacement therapy (RRT)--background of a developing German National Registry for RRT. QuaSi-Niere Task Group. Nephrol Dial Transplant. 1995;10(4):442-3. doi: 10.1093/ndt/10.4.442. No abstract available. PMID 7623980